CLINICAL TRIAL: NCT02533648
Title: Involvement of Reactive Oxygen Species Produced by the Xanthine Oxidase in Mitochondrial Alterations in Skeletal Muscle of Type 2 Diabetic Patients
Brief Title: Role of Allopurinol on Oxidative Stress and Mitochondrial Alterations in Skeletal Muscle of Diabetic Patients
Acronym: DIAXO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010.639
Record Dates: First submitted 2015-05-18; First posted 2015-08-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus, oxidative stress; insulin sensitivity; insulin resistance; mitochondrial dysfunction; skeletal muscle; xanthine oxidase; allopurinol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Mitochondrial Diseases | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): Allopurinol, experimental arms, type 2 diabetes subjects receive 2 capsules of allopurinol 150 mg daily for 3 month
  Interventions: Drug: 2 capsules of allopurinol 150 mg daily for 3 month
- Placebo (Placebo Comparator): Placebo, type 2 diabetes subjects receive 2 capsules of lactose (placebo) daily for 3 month
  Interventions: Drug: 2 capsules of lactose daily for 3 month

INTERVENTIONS:
Drug: 2 capsules of allopurinol 150 mg daily for 3 month — 2 capsules of allopurinol 150 mg daily for 3 month
  Arms: Allopurinol
Drug: 2 capsules of lactose daily for 3 month — 2 capsules of lactose daily for 3 month
  Arms: Placebo

SUMMARY:
Our recent data in mice have demonstrated a key role of xanthine oxidase in hyperglycemia-induced by Reactive oxygen species production, and a preventive role of allopurinol (inhibitor of xanthine oxidase) on the keeping of mitochondria number and structure, in skeletal muscle of diabetic mice. The investigators want to initiate a clinical trial in order to evaluate the efficacy of allopurinol on the improvement of mitochondrial alterations, oxidative capacities and insulin sensitivity, in skeletal muscle of type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI from 25 to 40 kg/m²
* Type 2 diabetes known for over one year but less than 10 years, treated with Oral anti-diabetic drugs or a Glucagon-like peptide-1 (GLP1-analog)
* well controlled hypertension (untreated or currently treated) with a systolic blood pressure of 95 to 140 mmHg and diastolic blood pressure of 45 to 90 mmHg and heart frequency of 40 to 100 per minute
* Recent HbA1c < 9 %
* Uricemia > 300 µmol/l
* For women : Menopausal or contraception
* Renal function as defined by glomerular filtration rate (GFR) ≥ 80 mL/min/1.73 m2

Exclusion Criteria:

* Tobacco ( more than 5 cigarettes)
* Excessive drinking
* Known pathology
* Hypersensitivity to allopurinol
* Treatment by anticoagulants, allopurinol, regular steroids or Nonsteroidal anti-inflammatory drug (NSAID), fibrate or insulin

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02-18 (Actual)

PRIMARY OUTCOMES:
muscle oxidative stress in diabetic patients | At 3 months of treatment
  muscular protein carbonylation level (unit: reactive carbonyl derivates, arbitrary unit) by Western blot (oxyblot kit from Chemicon) and pro et antioxidant genes expression (unit: mRNA levels normalized by housekeeping gene, arbitrary ratio) by real time polymerase chain reaction (RT-PCR)

SECONDARY OUTCOMES:
- plasmatic oxidative stress by dosing plasmaticmarkers: | At 3 months of treatment
  Dosing plasmatic malondialdéhyde, plasmatic H2O2, protein carbonylation of plasmatic protein and urinary isoprostans, and finally antioxidants (vitamins C and E, glutathione (unit: from µM to M)
alterations in mitochondrial structure of skeletal muscle with transmission electron microscopy | At 3 months of treatment
  Analysis of mitochondria area (in µm2) and density (in %)
mitochondrial density by measuring the ratio mitochondrial Deoxyribonucleic acid (mtDNA)/nuclear DNA by real-time polymerase chain reaction (PCR) in skeletal muscle | At 3 months of treatment
mitochondrial function | At 3 months of treatment
  Expression of genes implicated in mitochondrial action (messenger Ribonucleic acid (mRNA) levels by Reverse transcription polymerase chain reaction (RT-PCR) and proteins levels by Western Blot)(unit: arbitrary ratio relative to housekeeping gene/protein).
quantification of intramuscular lipids by histology (biopsy analysis) | At 3 months of treatment
  Staining Oil Red O evaluate the intramuscular lipid accumulation using the software ImageJ(unit: % of labelling by field).
sensitivity to insulin using a hyperinsulinemic euglycemic clamp | At 3 months of treatment
  sensitivity to insulin will be expressed as the glucose infusion rate (GIR)/insulinemia ratio.
uricemia and xanthine oxidase activity in sera and muscles(unit: mg/l for uricemia and mU/ml for XO activity) | At 3 months of treatment
  Plasma concentrations of uric acid will be measured before and after treatment to assess patient compliance . The reduction of xanthine oxidase activity in serum and muscle protein lysates will be measured using the kit " Amplex Red xanthine / xanthine oxidase assay kit" from Molecular Probes
Tolerance of the treatment measured by any adverse events during treatment and between each visit. | during the 3 months of treatment
  Any adverse events during treatment and between each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- CRNH Rhône Alpes, Lyon, France